CLINICAL TRIAL: NCT04617665
Title: Department of Anesthesiology, Fudan University Shanghai Cancer Center, Fudan University, Shanghai, China.
Brief Title: Effects of One-handed and Two-handed Mask Ventilation Techniques on Global and Regional Lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mask ventilation
Record Dates: First submitted 2020-10-25; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-handed mask ventilation (Other): For the one-handed mask ventilation, only one hand can be used to achieve the face mask seal. The left thumb and index finger form a ''C,'' providing anterior pressure over the mask, while the third, fourth, and fifth fingers form an ''E'' to lift the jaw.
  Interventions: Other: One-handed mask ventilation
- Two-handed mask ventilation (Other): For the two-handed mask ventilation, the provider's thumb and thenar eminence of each hand are held parallel, adjacent to the mask connector, and depress each side of the mask. The second through fifth digits wrap around and elevate the mandible to draw it anteriorly into the mask establishing both a jaw-thrust and chin-lift maneuver when appropriate.
  Interventions: Other: Two-handed mask ventilation

INTERVENTIONS:
Other: One-handed mask ventilation — Using one-handed mask ventilation techniques during induction of general anesthesia
  Arms: One-handed mask ventilation
Other: Two-handed mask ventilation — Using two-handed mask ventilation techniques during induction of general anesthesia
  Arms: Two-handed mask ventilation

SUMMARY:
Two-handed mask ventilation has been shown to provide higher tidal volume than one-handed mask ventilation. The effects of the two techniques on respiratory mechanics during induction of general anesthesia, however, still need to be determined.

DETAILED DESCRIPTION:
Mask positive pressure ventilation always causes the changes of respiratory mechanics such as ventral redistribution of regional ventilation, which impairs gas exchange. Two-handed mask ventilation has been shown to improve gas exchange by providing higher tidal volume than one-handed mask ventilation. We hypothesis that those higher tidal volume caused by two-handed mask ventilation would also improve the respiratory mechanics during induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery with general anesthesia
* American Society of Anesthesiologist (ASA) physical class of I-II.

Exclusion Criteria:

* acute and chronic respiratory disorders, including chronic obstructive
* pulmonary disease (COPD) and asthma;
* a history of lung surgery;
* exist risk of reflux and aspiration;
* patients requiring an awake intubation;
* facial and thoracic deformities;
* implants exist in the body, such as cardiac pacemakers;
* pregnant women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
global inhomogeneity (GI) | 8 weeks
  EIT images will be acquired by using the EIT monitor (Drager Medical Gmbh, Lubeck, Germany). And a software package (Electrical impedance tomography diag custom software provided by Drager Medical) will be used to quantitatively analyze the EIT data. 0% = homogenous

SECONDARY OUTCOMES:
centre of ventilation (CoV) | 8 weeks
  EIT images will be acquired by using the EIT monitor (Drager Medical Gmbh, Lubeck, Germany). And a software package (Electrical impedance tomography diag custom software provided by Drager Medical) will be used to quantitatively analyze the EIT data. 100% = entirely dorsal.
regional ventilation delay (RVD) | 8 weeks
  EIT images will be acquired by using the EIT monitor (Drager Medical Gmbh, Lubeck, Germany). And a software package (Electrical impedance tomography diag custom software provided by Drager Medical) will be used to quantitatively analyze the EIT data.
ventilation of regional lung ( %) | 8 weeks
  EIT images will be acquired by using the EIT monitor (Drager Medical Gmbh, Lubeck, Germany). And a software package (Electrical impedance tomography diag custom software provided by Drager Medical) will be used to quantitatively analyze the EIT data.
Expiratory tidal volume (TV) | 8 weeks
  Expiratory tidal volume will be recorded through the anesthesia machine.
PaO2/FiO2 | 8 weeks
  PaO2/FiO2 will be recorded through arterial blood gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: Yes
Data or documents can be obtained by contact the corresponding authors. Files can be emailed to anyone that concerned.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During the submission and after the acceptance.
Access Criteria: Anyone who is interested in or has questions in this study.